CLINICAL TRIAL: NCT02672137
Title: Knowledge Translation to Promote Evidence-based Medical Therapy in Acute Coronary Syndromes
Brief Title: Knowledge Translation for Patients With Acute Coronary Syndromes
Acronym: AMI-OPTIMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montreal General Hospital (Other)
Collaborators: Sanofi (Industry); Canadian Institutes of Health Research (CIHR) (Other Government); Fonds de la Recherche en Santé du Québec (Other Government)
Responsible Party: Principal Investigator, Thao Huynh, Cardiologist, associate professor of medicine, Montreal General Hospital
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: DIREG_L_04201
Record Dates: First submitted 2016-01-10; First posted 2016-02-03 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-01

CONDITIONS: Acute Coronary Syndromes
Keywords: myocardial infarction; knowledge transfer; acute coronary syndromes
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- knowledge translation (Experimental): knowledge translation 12-month multi-facet intensive knowledge translation measures that include: Community of practice, local gap analysis, opinion leaders, targeted interventions, performance feedback, reminders and local formation of ACS teams.
  Interventions: Behavioral: knowledge translation
- Usual care (No Intervention): no intervention

INTERVENTIONS:
Behavioral: knowledge translation — knowledge translation that include: Community of practice, local gap analysis, opinion leaders, targeted interventions, performance feedback, reminders and local formation of ACS teams.
  Arms: knowledge translation

SUMMARY:
Cluster randomized open-label experimental study multi-center of 24 hospitals to either knowledge translation vs usual care to improve care of patents hospitalized for acute coronary syndromes.

DETAILED DESCRIPTION:
The AMI-OPTIMA study was a cluster randomized controlled trial of 24 hospitals to one-year knowledge translation (KT) vs usual care. Prior to randomization, we reviewed charts of 100 consecutive acute coronary syndromes (ACS) patients at each participating hospital in 2009. During one year, hospitals randomized to KT completed: 1) revision of the most recent American Heart Association Guidelines of ACS management, 2) focus groups to identify and solve local care gaps, and 3)local champion team to promote evidence-based medical therapy (EBMT). At the end of 12-month of KT/usual care, we reviewed discharge prescriptions of 100 consecutive ACS patients at each participating hospital (year 2012).

EBMT was pre-defined as in-hospital anticoagulation and discharge prescription of dual anti-platelets, beta-blockers, statins, and angiotensin pathway modulating agents (for patients with impaired left ventricular systolic function). Refusal, impaired cognitive function, allergy or intolerance of patients to any of EBMT were considered valid reasons for withholding EBMT.

ELIGIBILITY:
Inclusion Criteria:Had a final discharge diagnosis of one of the following categories:

1. Myocardial infarction with ST-segment elevation
2. Myocardial infarction without ST-segment elevation
3. Unstable angina
4. Acute coronary syndromes -

Exclusion Criteria:

1. Non-atherosclerotic coronary artery disease (as confirmed by coronary angiograms or other non-invasive tests such as stress test, coronary CT-scan, nuclear scans)
2. Hospital stay of less than 48 hours -

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4604 (Actual)
Dates: Start 2010-01; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who received evidence-based medical therapy at hospital discharge (mean of 4 days) | at hospital discharge (average of 4 days)
  Evidence-based medical therapy is defined as aspirin,dual-antiplaquelets, beta-blockers, statins.

SECONDARY OUTCOMES:
Discharge prescription of individual evidence-based medical therapy: aspirin, dual antiplatelets, beta-blockers | at hospital discharge (average of 4 days)
  For each of the following medication: aspirin, dual anti-platelet, beta-blocker and statin, we calculated the proportion of patients who were prescribed the specific medication at discharge (as recorded on the discharge prescription).
Safety endpoints (mortality, reinfarction, strokes and bleeding outcomes (TIMI major and minor bleeds)) | in-hospital (average of 4 days)
  mortality, reinfarction, strokes and bleeding outcomes (TIMI major and minor bleeds)

CONTACTS AND LOCATIONS:
Overall Officials: thao huynh, md,msc,phd, Principal Investigator — Montreal General Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Huynh T, Kouz S, Afilalo M, Rinfret S, Schampaert E, Mansour S, Montigny M, Eisenberg MJ, Lauzon C, Dery JP, Nguyen M, L'Allier P, Harvey R, Boudreault C, Tardif JC. Knowledge Translation to improve prescription of evidence-based medical therapy for patients admitted with acute coronary syndromes: insights from the AMI-OPTIMA study. Journal of the American College of Cardiology.J Am Coll Cardiol. 2015;65(10_S).